CLINICAL TRIAL: NCT06013007
Title: Joint Inflation With Nominal-pressure and Stability Approach in Coronary Drug-Eluting Stent Optimization and Outcomes
Brief Title: Joint Inflation With Nominal-pressure and Stability Approach in DES Optimization
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zunyi Medical College (Other)
Responsible Party: Principal Investigator, Cai De Jin, MD, Principal Investigator, Zunyi Medical College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JINS
Record Dates: First submitted 2023-08-21; First posted 2023-08-28 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Acute Coronary Syndrome; De Novo Stenosis
Keywords: JINS; Intracoronary imaging; Stent optimization; Outcomes
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Intervention Model Description: Eligible patients will be implanted with DES by Joint Inflation with Nominal-pressure and Stability (JINS) approach, which is described as inflating a stent balloon with nominal-pressure without decay for at least 30 seconds.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JINS approach (Experimental): The JINS approach is described as inflating a stent balloon with nominal-pressure without decay for at least 30 seconds.
  Interventions: Procedure: ICI-guided JINS approach

INTERVENTIONS:
Procedure: ICI-guided JINS approach — OCT- or IVUS-guided JINS approach in DES implantation (DES types including Healing-Targeted SUPREME/Infinity Sirolimus-Eluting Stent, GuReater™ Sirolimus-Eluting Stent, XIENCE Alpine Everolimus-Eluting Stent, Promus PREMIER™ Everolimus-Eluting Stent, Resolute Integrity™ Zotarolimus-Eluting Stent, Firebird 2™ Sirolimus-Eluting Stent, Firekingfisher™ Sirolimus-Eluting Stent).

SUMMARY:
To achieve the stent optimization following "Keep It Simple and Safe" coronary intervention is recommended. A protocol of Joint Inflation with Nominal-pressure and Stability (JINS) approach in coronary drug-eluting stent (DES) implantation by intracoronary imaging (ICI) guidance could provide additional benefits in reducing unnecessary radiation exposure, and post-dilatation balloon angioplasty-related complications.

DETAILED DESCRIPTION:
Variable types of stent inflation protocol to achieve evidence and consensus-based coronary drug-eluting stent (DES) optimization could improve clinical outcomes. The investigators aim to evaluate whether the JINS approach could be adopted in Chinese daily practice.

The investigators will perform ICI (OCT or IVUS)-guided DES implantation in coronary de novo lesions by JINS protocol, described as inflating stent balloon with nominal-pressure (+1~2atm) without decay for at least 30 seconds.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute coronary syndrome (UA/NSTEMI/STEMI) plan to undergo OCT- or IVUS-guided DES implantation in de novo lesion.
* Patients provide written informed consent prior to enrollment.

Exclusion Criteria:

* Left main, ostial right coronary artery lesion.
* High thrombus burden at the index primary percutaneous coronary intervention.
* Active bleeding or bleeding diathesis, thrombocytopenia (platelet <100,000/mL), or hemoglobin <10 g/dL
* Hepatic dysfunction (serum liver enzyme>3 times the normal limit)
* Renal failure (eGFR <15 ml/min/1.73m2 or requiring dialysis)
* Life expectancy < 1 year

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2023-08-22 (Actual); Primary Completion 2025-08-22 (Estimated); Study Completion 2025-09-22 (Estimated)

PRIMARY OUTCOMES:
Stent optimization | At 24 hours
  To achieve the targets as follow: minimal stent area (MSA) >5.5 mm2 by IVUS or MSA >4.5mm2 by OCT, stent expansion >80% (MSA divided by average reference lumen area), no significant malapposition, no significant stent edge dissection, no significant tissue protrusion, and successful DES implantation without the occurrence of cardiac death, target vessel myocardial infarction, target lesion revascularization, acute stent thrombosis during the first 24 hours after an index procedure.

SECONDARY OUTCOMES:
Target vessel failure | At 12 months
  Composite of cardiac death, target vessel myocardial infarction, ischaemia-driven target vessel revascularization.

CONTACTS AND LOCATIONS:
Overall Officials: Cai De Jin, MD, Principal Investigator — Zunyi Medical College
Locations (1):
- Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou, China

REFERENCES:
- [Result] Hovasse T, Mylotte D, Garot P, Salvatella N, Morice MC, Chevalier B, Pichard A, Lefevre T. Duration of balloon inflation for optimal stent deployment: five seconds is not enough. Catheter Cardiovasc Interv. 2013 Feb;81(3):446-53. doi: 10.1002/ccd.23343. Epub 2012 Jan 10. PMID 22109977
- [Result] Ann SH, Chung JW, DE Jin C, Lee JH, Kim JM, Garg S, Shin ES. Better inflation time of stent balloon for second-generation drug-eluting stent expansion and apposition: an optical coherence tomography study. J Interv Cardiol. 2014 Apr;27(2):171-6. doi: 10.1111/joic.12096. Epub 2014 Mar 5. PMID 24593834
- [Result] Vallurupalli S, Kasula S, Kumar Agarwal S, Pothineni NVK, Abualsuod A, Hakeem A, Ahmed Z, Uretsky BF. A novel stent inflation protocol improves long-term outcomes compared with rapid inflation/deflation deployment method. Catheter Cardiovasc Interv. 2017 Aug 1;90(2):233-240. doi: 10.1002/ccd.26930. Epub 2017 Jan 23. PMID 28112479
- [Result] Raber L, Mintz GS, Koskinas KC, Johnson TW, Holm NR, Onuma Y, Radu MD, Joner M, Yu B, Jia H, Meneveau N, de la Torre Hernandez JM, Escaned J, Hill J, Prati F, Colombo A, di Mario C, Regar E, Capodanno D, Wijns W, Byrne RA, Guagliumi G; ESC Scientific Document Group. Clinical use of intracoronary imaging. Part 1: guidance and optimization of coronary interventions. An expert consensus document of the European Association of Percutaneous Cardiovascular Interventions. Eur Heart J. 2018 Sep 14;39(35):3281-3300. doi: 10.1093/eurheartj/ehy285. PMID 29790954